CLINICAL TRIAL: NCT02942238
Title: Standardization of Laparoscopic Surgery for Right Hemi Colon Cancer (SLRC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Minhua Zheng, professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ruijin-0002
Record Dates: First submitted 2016-10-20; First posted 2016-10-24 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Overall Survival; Postoperative Complications; Metastasis; Stage, Colon Cancer
Keywords: CME; Right hemi Colon cancer; D3; laparoscopy
MeSH Terms: conditions — Postoperative Complications; Neoplasm Metastasis; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Complete Mesocolic Excision (Experimental): the group underwent laparoscopic right hemicolectomy with CME. In complete mesocolic excision group (CME), the dissecting extent includes the lymphatic and fat tissues surrounding the root of ascending mesocolon, which situated on the surface of superior mesenteric vein, and the root of right half of transverse mesocolon, which situated on the surface of pancreas neck.
  Interventions: Procedure: CME
- D3 lymph node dissection (Active Comparator): the group underwent laparoscopic right hemicolectomy with D3 lymph node dissection. In D3 lymph node dissection group(D3), the lymph node dissection is based on ligating the supplying vessels close to the right-side of superior mesenteric vein and clean up the surrounding lymph node and adipose tissue. No.6 lymph node should be dissected in this group.
  Interventions: Procedure: D3

INTERVENTIONS:
Procedure: CME — the group underwent laparoscopic right hemicolectomy with CME. In CME group, in addition to D2 dissection, the whole mesocolon, from ascending colon to right half transverse colon, as well as the central lymph nodes should be entirely removed.
  Intervention: Procedure: Complete mesocolic excision (CME)
  Arms: Complete Mesocolic Excision
Procedure: D3 — the group underwent laparoscopic right hemicolectomy with D3 lymph node dissection. In D3 group, the mesocolon should be removed and the dissection involves the paracolon and intermediate lymph nodes,including No.6 lymph node, which along the feeding vessels.
  Intervention: Procedure: D3 radical operation
  Arms: D3 lymph node dissection

SUMMARY:
To standardize the surgery for advanced right hemi colon cancer with laparoscopy and investigate whether extended lymphadenectomy (CME) could improve disease-free survival in patients with right colon cancer, compared with D3 radical operation in laparoscopic colectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suitable for curative surgery 18-75years old
2. Qualitative diagnosis: a pathological diagnosis of adenocarcinoma;
3. Localization diagnosis: the tumor located between the cecum and the right 1/3 of transverse colon;
4. Enhanced CT scan of chest, abdominal and pelvic cavity: assessment of tumor stage is T stage 1-4 and N stage 0-2; there is no distant metastasis.
5. Informed consent

Exclusion Criteria:

1. Simultaneous or simultaneous multiple primary colorectal cancer;
2. Preoperative imaging examination results show: (1) Tumor involves the surrounding organs and combined organ resection need to be done; (2)distant metastasis; (3)unable to perform R0 resection;
3. History of any other malignant tumor in recent 5 years;
4. Patients need emergency operation;
5. Not suitable for laparoscopic surgery;
6. Women during Pregnancy or breast feeding period;
7. Informed consent refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years

SECONDARY OUTCOMES:
The rate of postoperative complications and mortality | 30 days
3 years overall survival | 3 years
The rate of local and distant recurrence | 3 years
The accuracy of preoperative staging with CT | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Minhua Zheng, PhD, Study Director — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ostenfeld EB, Erichsen R, Iversen LH, Gandrup P, Norgaard M, Jacobsen J. Survival of patients with colon and rectal cancer in central and northern Denmark, 1998-2009. Clin Epidemiol. 2011;3 Suppl 1(Suppl 1):27-34. doi: 10.2147/CLEP.S20617. Epub 2011 Jul 21. PMID 21814467
- [Result] Laparoscopically assisted colectomy is as safe and effective as open colectomy in people with colon cancer Abstracted from: Nelson H, Sargent D, Wieand HS, et al; for the Clinical Outcomes of Surgical Therapy Study Group. A comparison of laparoscopically assisted and open colectomy for colon cancer. N Engl J Med 2004; 350: 2050-2059. Cancer Treat Rev. 2004 Dec;30(8):707-9. doi: 10.1016/j.ctrv.2004.09.001. No abstract available. PMID 15541580
- [Result] Kitano S, Inomata M, Sato A, Yoshimura K, Moriya Y; Japan Clinical Oncology Group Study. Randomized controlled trial to evaluate laparoscopic surgery for colorectal cancer: Japan Clinical Oncology Group Study JCOG 0404. Jpn J Clin Oncol. 2005 Aug;35(8):475-7. doi: 10.1093/jjco/hyi124. Epub 2005 Jul 8. PMID 16006574
- [Result] Guillou PJ, Quirke P, Thorpe H, Walker J, Jayne DG, Smith AM, Heath RM, Brown JM; MRC CLASICC trial group. Short-term endpoints of conventional versus laparoscopic-assisted surgery in patients with colorectal cancer (MRC CLASICC trial): multicentre, randomised controlled trial. Lancet. 2005 May 14-20;365(9472):1718-26. doi: 10.1016/S0140-6736(05)66545-2. PMID 15894098
- [Result] Engstrom PF, Arnoletti JP, Benson AB 3rd, Chen YJ, Choti MA, Cooper HS, Covey A, Dilawari RA, Early DS, Enzinger PC, Fakih MG, Fleshman J Jr, Fuchs C, Grem JL, Kiel K, Knol JA, Leong LA, Lin E, Mulcahy MF, Rao S, Ryan DP, Saltz L, Shibata D, Skibber JM, Sofocleous C, Thomas J, Venook AP, Willett C; National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: colon cancer. J Natl Compr Canc Netw. 2009 Sep;7(8):778-831. doi: 10.6004/jnccn.2009.0056. No abstract available. PMID 19755046
- [Result] West NP, Kobayashi H, Takahashi K, Perrakis A, Weber K, Hohenberger W, Sugihara K, Quirke P. Understanding optimal colonic cancer surgery: comparison of Japanese D3 resection and European complete mesocolic excision with central vascular ligation. J Clin Oncol. 2012 May 20;30(15):1763-9. doi: 10.1200/JCO.2011.38.3992. Epub 2012 Apr 2. PMID 22473170
- [Result] Kobayashi H, West NP, Takahashi K, Perrakis A, Weber K, Hohenberger W, Quirke P, Sugihara K. Quality of surgery for stage III colon cancer: comparison between England, Germany, and Japan. Ann Surg Oncol. 2014 Jun;21 Suppl 3:S398-404. doi: 10.1245/s10434-014-3578-9. Epub 2014 Feb 25. PMID 24566862
- [Result] Bertelsen CA, Neuenschwander AU, Jansen JE, Wilhelmsen M, Kirkegaard-Klitbo A, Tenma JR, Bols B, Ingeholm P, Rasmussen LA, Jepsen LV, Iversen ER, Kristensen B, Gogenur I; Danish Colorectal Cancer Group. Disease-free survival after complete mesocolic excision compared with conventional colon cancer surgery: a retrospective, population-based study. Lancet Oncol. 2015 Feb;16(2):161-8. doi: 10.1016/S1470-2045(14)71168-4. Epub 2014 Dec 31. PMID 25555421
- [Result] Eiholm S, Ovesen H. Total mesocolic excision versus traditional resection in right-sided colon cancer - method and increased lymph node harvest. Dan Med Bull. 2010 Dec;57(12):A4224. PMID 21122462